CLINICAL TRIAL: NCT03523065
Title: The Chinese Parkinson's Disease With GBA Variants Registry
Brief Title: Chinese PD-GBA Registry
Status: Recruiting | Type: Observational
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: CPD-GBAR
Record Dates: First submitted 2018-05-01; First posted 2018-05-14 (Actual); Last update posted 2018-05-29 (Actual); Status verified 2018-04

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the Chinese Parkinson's disease with GBA variants Registry (CPD-GBAR) is to develop a database of patients of Parkinson's disease with Glucocerebrosidase (GBA) gene variants in mainland China.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is the second most common disorder among neurodegenerative diseases. GBA gene variants such as L444P can influence the risk of developing PD and these variants have the greatest impact on PD susceptibility among all the PD related gene variants yet discovered. The investigators aim to establish a database of PD with GBA variants and characterize the clinical manifestation of these patients in mainland China.

Method:

1. Peripheral blood from patients has been tested to have GBA gene variants.
2. Clinical manifestation will be measured by scales and neurological tests. Standard scales include: Unified Parkinson's Disease Rating Scale(UPDRS), Hoehn-Yahr stages, Non-Motor Symptoms Scale (NMSS), mini-mental state examination (MMSE), Parkinson disease sleep scales (PDSS), Rapid Eye Movement Sleep Behaviour Disorder Questionnaire(RBDQ-HK), Epworth Sleepiness Scale (ESS), Rome III functional constipation scale, the Scale for Outcomes in PD for Autonomic Symptoms (SCOPA-AUT), Parkinson Fatigue Scale (PFS), Cambridge-Hopkins Restless Legs Syndrome questionnaire (CHRLSq), Hyposmia rating scale(HRS), Hamilton depression scale, the 39-item Parkinson's Disease Questionnaire(PDQ-39), Freezing of gait scale(FOG), dyskinesia related scales, Wearing-off scale(WO).
3. The investigators will also exam the blood biomarkers of PD such as uric acid and peripheral inflammatory markers.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with PD by the United Kingdom Parkinson's Disease Society Brain Bank clinical diagnostic criteria or other standard criteria; PD patients detected with GBA gene variants.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: PD patients with GBA gene variants
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Database of Parkinson's disease with GBA variants | 10 years
  Establish the database of Parkinson's disease with GBA variants in mainland China.
Clinical feature | 10 years
  Characterize the clinical feature of PD patients with GBA variants

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangya Hospital of Central South University, Changsha, Hunan, China

REFERENCES:
- [Background] Zhang Y, Shu L, Sun Q, Zhou X, Pan H, Guo J, Tang B. Integrated Genetic Analysis of Racial Differences of Common GBA Variants in Parkinson's Disease: A Meta-Analysis. Front Mol Neurosci. 2018 Feb 15;11:43. doi: 10.3389/fnmol.2018.00043. eCollection 2018. PMID 29527153
- [Result] Sun QY, Guo JF, Wang L, Yu RH, Zuo X, Yao LY, Pan Q, Xia K, Tang BS. Glucocerebrosidase gene L444P mutation is a risk factor for Parkinson's disease in Chinese population. Mov Disord. 2010 Jun 15;25(8):1005-11. doi: 10.1002/mds.23009. PMID 20131388
- [Result] Guo JF, Li K, Yu RL, Sun QY, Wang L, Yao LY, Hu YC, Lv ZY, Luo LZ, Shen L, Jiang H, Yan XX, Pan Q, Xia K, Tang BS. Polygenic determinants of Parkinson's disease in a Chinese population. Neurobiol Aging. 2015 Apr;36(4):1765.e1-1765.e6. doi: 10.1016/j.neurobiolaging.2014.12.030. Epub 2015 Jan 6. PMID 25623333
- [Result] Zhang Y, Sun QY, Zhao YW, Shu L, Guo JF, Xu Q, Yan XX, Tang BS. Effect of GBA Mutations on Phenotype of Parkinson's Disease: A Study on Chinese Population and a Meta-Analysis. Parkinsons Dis. 2015;2015:916971. doi: 10.1155/2015/916971. Epub 2015 Sep 2. PMID 26421210
- [Result] Fan K, Tang BS, Wang YQ, Kang JF, Li K, Liu ZH, Sun QY, Xu Q, Yan XX, Guo JF. The GBA, DYRK1A and MS4A6A polymorphisms influence the age at onset of Chinese Parkinson patients. Neurosci Lett. 2016 May 16;621:133-136. doi: 10.1016/j.neulet.2016.04.014. Epub 2016 Apr 13. PMID 27085534